CLINICAL TRIAL: NCT02007642
Title: Performance Assessment of High Throughput Sequencing for the Detection of Pathogens in Immunocompromised Patients With Suspected Infectious Disease.
Brief Title: Evaluation of High Throughput Sequencing for Screening of Pathogens in Immunocompromised Patients With Suspected Infectious Disease.
Acronym: PATHOQUEST1
Status: Completed | Type: Observational
Sponsor: Pathoquest (Industry)
Collaborators: Imagine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PTQCT01-2013
Record Dates: First submitted 2013-11-29; First posted 2013-12-11 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2013-10

CONDITIONS: Immunodeficiency and Suspected Infection
MeSH Terms: conditions — Immunologic Deficiency Syndromes | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA sample by patient
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No study treatment
  Interventions: Procedure: Blood sampling / Body fluid sampling

INTERVENTIONS:
Procedure: Blood sampling / Body fluid sampling — During the hospitalization of the patient, when a sampling is done for classic follow-up and diagnosis, additionnal blood sampling will be done, for the PATHOQUEST method.
  Other body fluids might be taken (if the sampling is done for the classic follow-up), such as cerebrospinal fluid, ascite...

SUMMARY:
The study patients are patients suffering from primary or secondary immunodeficiencies investigated in the Hospital Necker for a suspected infectious disease.

The study purpose is to assess the performance of a High Throughput Sequencing method, the PATHOQUEST method (from sample preparation to bio informatic analysis), versus the classic diagnostic approach.

The study will evaluate the capacity of the PATHOQUEST method to detect pathogens responsible for an infectious disease episode and will also evaluate the delay of obtention of results compared to the classic diagnostic approach.

ELIGIBILITY:
Summary of inclusion criteria:

1. Primary or secondary immunodeficiencies defined by

   * Solid organ transplantation and immunosuppressive drug
   * Recent chemotherapy
   * Hematopoïetic Stem Cells transplantation
   * Primary immune deficiency
   * Auto-immune disease
   * HIV infection
2. Infection suspicion
3. Microbiological investigation
4. Adult or child above 1 year
5. Hospitalization at Necker-Enfants malades hospital
6. Registration to Healthcare organism
7. ICF signature

Summary of exclusion criteria:

1. Obvious diagnosis following clinical examination
2. Participation in a clinical trial for a new drug
3. People under legal guardianship
4. People unable to fulfil the required medical follow-up

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Immunocompromised patients hospitalized for a suspected infectious disease
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Identification of pathogens responsible for the infection | 1 year
  The primary outcome will assess the number of diagnostics obtained by the PATHOQUEST method and classic diagnostic approach.

SECONDARY OUTCOMES:
Delay of obtention of diagnostic | 1 year
  The delay of obtention of results will be compared to determine which approach allows an earlier diagnosis.
Economic impact of the PATHOQUEST method | 1 year
  Comparison of the cost of the classic diagnostic approach and PATHOQUEST method, including cost of the hospital stay, microbiological tests performed, empirical anti-infectious drugs prescribed.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Lecuit, Pr, Principal Investigator — marc.lecuit@nck.aphp.fr
Locations (2):
- France (2):
  - Hôpital Européen Georges Pompidou, Paris
  - Hopital Necker - Enfants malades, Paris, Île-de-France Region